CLINICAL TRIAL: NCT03874715
Title: Randomized, Open Label, Parallel-group Study Comparing the Pharmacokinetics and Immunogenicity of Alternating Use of SAR341402 and NovoLog® Versus Continuous Use of NovoLog in Participants With Type 1 Diabetes Mellitus Also Using Insulin Glargine
Brief Title: Comparison of SAR341402 to NovoLog in Adult Patients With Type 1 Diabetes Mellitus Also Using Insulin Glargine
Acronym: GEMELLI X
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC15178; U1111-1197-7811 (Other: UTN); 136342 (Other: IND)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Switching: NovoLog/SAR341402 (Experimental): Participants self-administered subcutaneous (SC) injection daily prior to the start of a meal during the 16-week treatment period, starting with NovoLog (100 units per milliliters [U/mL]) for the first 4 weeks, then SAR341402 (100 U/mL) for 4 weeks, followed by NovoLog (at same dose) for 4 weeks and then SAR341402 (at same dose) for the last 4 weeks on top of mandatory background therapy with Lantus (Insulin glargine, 100 U/mL) as basal insulin.
  Interventions: Drug: Insulin Aspart SAR341402; Drug: Insulin Aspart; Drug: Insulin glargine U100
- Non-Switching: NovoLog (Active Comparator): Participants self-administered SC injection of NovoLog (100 U/mL) daily prior to the start of a meal during the 16-week treatment period on top of mandatory background therapy with Lantus (Insulin glargine, 100 U/mL) as basal insulin.
  Interventions: Drug: Insulin Aspart; Drug: Insulin glargine U100

INTERVENTIONS:
Drug: Insulin Aspart SAR341402 — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous
  Arms: Switching: NovoLog/SAR341402
Drug: Insulin Aspart — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous
  Other Names: NovoLog
Drug: Insulin glargine U100 — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous
  Other Names: Lantus

SUMMARY:
Primary Objective:

To demonstrate similarity in pharmacokinetics (PK) of SAR341402 and NovoLog after 4x4-week periods of alternating administration of SAR341402 and NovoLog compared to 16-week continuous use of NovoLog in participants with Type 1 diabetes mellitus (T1DM) also using insulin glargine.

Secondary Objectives:

* To compare the effects of alternating administration of SAR341402 and NovoLog with continuous use of NovoLog on immunogenicity.
* To evaluate the safety of alternating administration of SAR341402 and NovoLog versus continuous use of NovoLog.
* To compare other PK parameters between the two treatment arms (alternating administration of SAR341402 and NovoLog and continuous use of NovoLog).

DETAILED DESCRIPTION:
The study duration per participant was less than 19 weeks (for participants who did not require the run-in period) and less than 31 weeks (for participants who require the run-in period).

ELIGIBILITY:
Inclusion criteria:

* Participants with T1DM.
* Participants on continuous insulin treatment for at least 12 months prior to screening.
* Participants exclusively on a multiple (greater than or equal to 3) daily injection insulin analogue regimen using:

  * NovoLog as mealtime insulin for at least 12 weeks prior to screening and
  * Insulin glargine (100 units per milliliter [U/mL]) as basal insulin for at least 12 weeks prior to screening. Note: Participants not meeting this criterion could also qualify, provided that they completed the run-in period during which NovoLog and Lantus was administered so that, at the time of randomization, the participants had been on NovoLog and insulin glargine (100 U/mL) for at least 12 weeks (including any potential pre-screening administration).
* Glycated hemoglobin (HbA1c) less than or equal to 10 percent (%) (85.79 millimoles per mole) at screening.
* Body mass index less than or equal to 35 kilograms per meter square (kg/m^2) at screening.

Exclusion criteria:

* Pancreatectomy and/or islet cell transplantation.
* Clinically significant laboratory findings, as defined by the protocol.
* Known presence of factors that interfered with the HbA1c measurement.
* History of severe hypoglycemia required emergency room admission or hospitalization within 3 months prior to screening.
* Hospitalization for recurrent diabetic ketoacidosis within 3 months prior to screening.
* Retinopathy or maculopathy with one of the following treatments, either recent (within 3 months of screening) or planned: intravitreal injections or laser or vitrectomy surgery.
* Use of glucose lowering treatments other than the multiple dose injections and basal insulin regimen (including use of insulin pump therapy), within 12 weeks prior to screening.
* Participants had received systemic glucocorticoids for one week or more within 3 months prior to screening (topical, nasal spray, inhaled or intra-articular applications are allowed).
* Participants had received systemic immunosuppressive agents within 6 months prior to screening.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (33):
- United States (33):
  - Investigational Site Number 8400014, Concord, California
  - Investigational Site Number 8400001, Temecula, California
  - Investigational Site Number 8400015, Ventura, California
  - Investigational Site Number 8400010, Aurora, Colorado
  - Investigational Site Number 8400029, Waterbury, Connecticut
  - Investigational Site Number 8400038, Doral, Florida
  - Investigational Site Number 8400030, Miami, Florida
  - Investigational Site Number 8400032, New Port Richey, Florida
  - Investigational Site Number 8400026, Ocoee, Florida
  - Investigational Site Number 8400033, Palm Harbor, Florida
  - Investigational Site Number 8400012, Atlanta, Georgia
  - Investigational Site Number 8400005, Columbus, Georgia
  - Investigational Site Number 8400009, Roswell, Georgia
  - Investigational Site Number 8400019, Crystal Lake, Illinois
  - Investigational Site Number 8400028, Des Moines, Iowa
  - Investigational Site Number 8400018, Lexington, Kentucky
  - Investigational Site Number 8400023, Baltimore, Maryland
  - Investigational Site Number 8400003, Rockville, Maryland
  - Investigational Site Number 8400013, Waltham, Massachusetts
  - Investigational Site Number 8400004, Flint, Michigan
  - Investigational Site Number 8400021, Kansas City, Missouri
  - Investigational Site Number 8400031, Washington, Missouri
  - Investigational Site Number 8400036, Omaha, Nebraska
  - Investigational Site Number 8400017, Las Vegas, Nevada
  - Investigational Site Number 8400007, New York, New York
  - Investigational Site Number 8400006, Morehead City, North Carolina
  - Investigational Site Number 8400035, Rocky Mount, North Carolina
  - Investigational Site Number 8400034, Jefferson City, Tennessee
  - Investigational Site Number 8400040, Dallas, Texas
  - Investigational Site Number 8400042, El Paso, Texas
  - Investigational Site Number 8400027, Houston, Texas
  - Investigational Site Number 8400016, Mesquite, Texas
  - Investigational Site Number 8400041, Waco, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Shah VN, Al-Karadsheh A, Barnes C, Mandry J, Nakhle S, Wernicke-Panten K, Kramer D, Schmider W, Pierre S, Teichert L, Rotthaeuser B, Mukherjee B, Bailey TS. Pharmacokinetic similarity of switching SAR341402 insulin aspart biosimilar and NovoLog insulin aspart versus continuous use of NovoLog in adults with type 1 diabetes: The GEMELLI X trial. Diabetes Obes Metab. 2024 Feb;26(2):540-547. doi: 10.1111/dom.15341. Epub 2023 Oct 25. PMID 37880868
- [Result] Shah VN, Al-Karadsheh A, Barnes C, Mandry J, Nakhle S, Wernicke-Panten K, Kramer D, Schmider W, Pierre S, Teichert L, Rotthaeuser B, Mukherjee B, Bailey TS. Safety and Efficacy of Switching SAR341402 Insulin Aspart and Originator Insulin Aspart vs Continuous Use of Originator Insulin Aspart in Adults With Type 1 Diabetes: The GEMELLI X Trial. J Diabetes Sci Technol. 2025 Jul;19(4):1051-1059. doi: 10.1177/19322968241232709. Epub 2024 Feb 29. PMID 38420944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 31 active sites in the United States. A total of 279 participants were screened from 11 March 2019 to 30 Oct 2019, out of which 210 participants were randomized. Participants were randomized in 1:1 ratio to "switching arm" (NovoLog/SAR341402) and "non-switching arm" (NovoLog). Randomization was stratified by glycated hemoglobin A1c (HbA1c) (less than [<] 8.0 percent [%] and greater than or equal to [>=] 8.0%) obtained at screening visit.
Pre-assignment Details: Participants not treated with NovoLog and insulin glargine (100 units per milliliter [U/mL] for at least 12 weeks prior to screening, completed a mandatory run-in period of up to 12-weeks and were administered NovoLog and Lantus. Run-in period duration was considered as a sufficient duration to ensure that, at the time of randomization, all the participants had received NovoLog and insulin glargine (100 U/mL) for at least 12 weeks.
Groups:
- Switching: NovoLog/SAR341402: Participants self-administered subcutaneous (SC) injection daily prior to the start of a meal during the 16-week treatment period, starting with NovoLog (100 U/mL) for the first 4 weeks, then SAR341402 (100 U/mL) for 4 weeks, followed by NovoLog (at same dose) for 4 weeks and then SAR341402 (at same dose) for the last 4 weeks on top of mandatory background therapy with Lantus (Insulin glargine, 100 U/mL) as basal insulin.
Period: Overall Study
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Started | 104 | 106
Treated | 104 | 106
Safety Population (Safety population included all randomized participants who received at least one dose of investigational medicinal product (IMP) and analyzed according to the treatment actually received.) | 99 | 111 (Five participants randomized to switching arm discontinued IMP during the first treatment of NovoLog before switching to SAR341402, thus included in the non-switching arm for the safety analysis.)
Anti-insulin Antibody (AIA) Population (AIA population included all participants who received at least one dose of IMP and with at least one AIA sample available for analysis, and were analyzed according to the treatment actually received) | 98 | 107 (Five participants randomized to switching arm discontinued IMP during the first treatment of NovoLog before switching to SAR341402, thus included in the non-switching arm for the AIA evaluations.)
Completed | 95 | 105
Not Completed | 9 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Poor compliance to protocol | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other-unspecified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population which included all participants who had a treatment kit number allocated and recorded in the interactive response technology (IRT) database, regardless of whether the treatment kit was used.
Groups:
- Switching: NovoLog/SAR341402: Participants self-administered SC injection daily prior to the start of a meal during the 16-week treatment period, starting with NovoLog (100 U/mL) for the first 4 weeks, then SAR341402 (100 U/mL) for 4 weeks, followed by NovoLog (at same dose) for 4 weeks and then SAR341402 (at same dose) for the last 4 weeks on top of mandatory background therapy with Lantus (Insulin glargine, 100 U/mL) as basal insulin.
- Total: Total of all reporting groups
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog | Total
Number analyzed (Participants) | 104 | 106 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (16.2) | 44.3 (15.8) | 44.1 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 84
  Male | 60 | 66 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 91 | 90 | 181
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve From Time Zero to Last Measurable Timepoint (AUClast) of Insulin Aspart Following Administration of Either SAR341402 (Switching Arm) or NovoLog (Non-switching Arm)
Description: AUClast was defined as area under the plasma concentration versus time curve from time zero to last measurable timepoint. Insulin aspart was the active ingredient of SAR341402 and NovoLog.
Time Frame: 0 hour (hr)(Pre-dose), 10, 20, 30, 40 & 50 minutes (min), 1hr, 1hr-10, 20, 30, 40 & 50min, 2hr, 2hr-15, 30 & 45min, 3hr, 3hr-15, 30 & 45min, 4hr, 4hr-20 & 40min, 5hr, 5hr-20 & 40min, 6hr, 6hr-30min, 7hr, 7hr-30min & 8hr post-dose on Day 112
Population: Analysis was performed on PK population which included all randomized participants without deviation that could significantly impact the PK analysis and for whom PK data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: picograms*hour per milliliter (pg*h/mL)
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Number analyzed (Participants) | 58 | 71
picograms*hour per milliliter (pg*h/mL) | 8960 (18300) | 7190 (6530)

2. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve (AUC) of Insulin Aspart Following Administration of Either SAR341402 (Switching Arm) or NovoLog (Non-switching Arm)
Description: AUC was defined as area under the concentration versus time curve. Insulin aspart is the active ingredient of SAR341402 and NovoLog.
Time Frame: 0 hr (pre-dose), 10, 20, 30, 40 & 50 min, 1 hr, 1 hr-10, 20, 30, 40 & 50 min, 2 hr, 2 hr-15, 30 & 45 min, 3 hr, 3 hr-15, 30 & 45 min, 4 hr, 4 hr-20 & 40 min, 5 hr, 5 hr-20 & 40 min, 6 hr, 6 hr-30 min, 7 hr, 7 hr-30 min & 8 hr post-dose on Day 112
Population: Analysis was performed on PK population. Here, "overall number of participants analyzed" = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Number analyzed (Participants) | 55 | 66
pg*h/mL | 6720 (3700) | 7260 (6370)

3. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of Insulin Aspart Following Administration of Either SAR341402 (Switching Arm) or NovoLog (Non-switching Arm)
Description: Cmax was defined as the maximum observed plasma concentration. Insulin aspart is the active ingredient of SAR341402 and NovoLog.
Time Frame: 0 hr (pre-dose), 10, 20, 30, 40 & 50 min, 1 hr, 1 hr-10, 20, 30, 40 & 50 min, 2 hr, 2hr-15, 30 & 45 min, 3 hr, 3 hr-15, 30 & 45 min, 4 hr, 4 hr-20 & 40 min, 5 hr, 5 hr-20 & 40 min, 6 hr, 6 hr-30 min, 7 hr, 7 hr-30 min & 8 hr post-dose on Day 112
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Number analyzed (Participants) | 58 | 71
picograms per milliliter (pg/mL) | 11800 (65600) | 3330 (8850)

4. Secondary Outcome: Number of Participants With Treatment-emergent Anti-Insulin Aspart Antibodies (AIAs)
Description: AIA was categorized as: treatment-induced AIA, treatment-boosted AIA, and treatment-emergent AIA. Treatment-induced AIAs: participants who developed AIA following investigational medicinal product (IMP) administration (participants with at least one positive AIA sample at any time during on-treatment period, in those participants without pre-existing AIA or with missing Baseline sample). Treatment-boosted AIAs: participants with pre-existing AIAs that were boosted to a significant higher titer following IMP administration (participants with at least one AIA sample with at least a 4-fold increase in titers compared to Baseline value at any time during on-treatment period, in those participants with pre-existing AIA). Participants with treatment-emergent AIA were defined as participants with treatment-induced, or treatment-boosted AIAs. On-treatment period was defined as the time from the first injection of IMP up to the last injection of IMP + 1 day.
Time Frame: From first injection of IMP (Day 1) up to 1 day after the last injection of IMP (i.e., up to Day 113)
Population: Analyzed on AIA population which included all randomized participants who received at least one dose of IMP and with at least one AIA sample available for analysis and were analyzed according to treatment actually received. Here, "number analyzed" = participants with available data for each specified category. Five participants randomized to switching arm discontinued IMP during first treatment of NovoLog before switching to SAR341402, thus included in non-switching arm for the AIA evaluations.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Number analyzed (Participants) | 98 | 107
Participants
  Treatment-emergent AIA | 8 | 11
  Treatment-boosted AIA: number analyzed (Participants) | 42 | 43
  Treatment-boosted AIA | 0 | 1
  Treatment-induced AIA: number analyzed (Participants) | 56 | 64
  Treatment-induced AIA | 8 | 10

5. Secondary Outcome: Number of Participants With at Least One Hypoglycemic Event
Description: Severe hypoglycemia: event in which participant required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions, because participant was not capable of helping self. Documented symptomatic hypoglycemia: event in which typical symptoms of hypoglycemia (SOH) were accompanied by measured plasma glucose concentration (PGC) less than or equal to (<=) 3.9 millimoles per liter (mmol/L)(<70 milligrams per deciliter [mg/dL]) or <3.0 mmol/L(<54 mg/dL). Asymptomatic hypoglycemia: event without SOH and with measured PGC of <=3.9 mmol/L (<70 mg/dL) or <3.0 mmol/L (<54 mg/dL). Probable symptomatic hypoglycemia: event with SOH not accompanied by plasma glucose determination but was presumably caused by PGC <=3.9 mmol/L (70 mg/dL). Relative hypoglycemia: event with SOH but with measured PGC greater than (>) 3.9 mmol/L (70 mg/dL).
Time Frame: From first injection of IMP (Day 1) up to 1 day after the last injection of IMP (i.e., up to Day 113)
Population: Analysis was performed on safety population which included all randomized participants who received at least one dose of IMP and analyzed according to the treatment actually received. Five participants randomized to switching arm discontinued IMP during the first treatment of NovoLog before switching to SAR341402, thus included in the non-switching arm for the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Number analyzed (Participants) | 99 | 111
Participants
  Any hypoglycemia | 95 | 105
  Severe hypoglycemia | 6 | 4
  Documented symptomatic hypoglycemia <=3.9 mmol/L | 89 | 98
  Documented symptomatic hypoglycemia < 3.0 mmol/L | 78 | 90
  Asymptomatic hypoglycemia <= 3.9 mmol/L | 69 | 68
  Asymptomatic hypoglycemia < 3.0 mmol/L | 48 | 44
  Probable symptomatic hypoglycemia | 8 | 9
  Relative hypoglycemia | 3 | 2

6. Secondary Outcome: Number of Hypoglycemic Events Per Participant-year
Description: Number of hypoglycemia events (any, severe, documented [both threshold], asymptomatic [both threshold], probable symptomatic and relative) per participant-year of exposure were reported. Severe hypoglycemia: event in which participant required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions, because participant wasn't capable of helping self. Documented symptomatic hypoglycemia: event in which typical SOH were accompanied by measured PGC of <=3.9 mmol/L (<70 mg/dL) or <3.0 mmol/L(<54 mg/dL). Asymptomatic hypoglycemia: event without SOH and measured PGC of <=3.9 mmol/L (<70 mg/dL) or <3.0 mmol/L(<54 mg/dL). Probable symptomatic hypoglycemia: event with SOH not accompanied by plasma glucose determination but was presumably caused by PGC <=3.9 mmol/L (70 mg/dL). Relative hypoglycemia: event with SOH but with measured PGC >3.9 mmol/L (70 mg/dL).
Time Frame: From first injection of IMP (Day 1) up to 1 day after the last injection of IMP (i.e., up to Day 113)
Population: Analysis was performed on safety population. Five participants randomized to switching arm discontinued IMP during the first treatment of NovoLog before switching to SAR341402, thus included in the non-switching arm for the safety analysis.
Measure: Number; unit: events per participant-year
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Number analyzed (Participants) | 99 | 111
events per participant-year
  Any hypoglycemia | 103.18 | 97.09
  Severe hypoglycemia | 0.76 | 0.38
  Documented symptomatic hypoglycemia <= 3.9 mmol/L | 64.29 | 63.54
  Documented symptomatic hypoglycemia < 3.0 mmol/L | 27.72 | 25.70
  Asymptomatic hypoglycemia <= 3.9 mmol/L | 37.33 | 32.25
  Asymptomatic hypoglycemia < 3.0 mmol/L | 9.11 | 7.03
  Probable symptomatic hypoglycemia | 0.70 | 0.81
  Relative hypoglycemia | 0.09 | 0.12

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) were defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/ incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the on-treatment period (from first injection of IMP up to 1 day after the last injection of IMP).
Time Frame: From first injection of IMP (Day 1) up to 1 day after the last injection of IMP (i.e., up to Day 113)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Number analyzed (Participants) | 99 | 111
Participants
  Any TEAEs | 25 | 47
  Any TESAEs | 5 | 5

8. Secondary Outcome: Pharmacokinetics: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Insulin Aspart Following Administration of Either SAR341402 (Switching Arm) or NovoLog (Non-switching Arm)
Description: Tmax was defined as the time taken to reach the maximum observed plasma concentration. Insulin aspart is the active ingredient of SAR341402 and NovoLog.
Time Frame: as for outcome 3
Population: Analysis was performed on PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
Number analyzed (Participants) | 58 | 71
hours | 1.33 [0.30 to 3.25] | 1.00 [0.37 to 3.13]

ADVERSE EVENTS:
Time Frame: From first injection of IMP (Day 1) up to 1 day after the last injection of IMP (i.e., up to Day 113)
Description: Analysis was performed on safety population. Five participants randomized to switching arm discontinued IMP during the first treatment of NovoLog before switching to SAR341402, thus included in the non-switching arm for the safety analysis.
Arm/Group | Switching: NovoLog/SAR341402 | Non-switching: NovoLog
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/111
Serious Adverse Events (participants affected / at risk) | 5/99 | 5/111
Other Adverse Events (participants affected / at risk) | 3/99 | 12/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switching: NovoLog/SAR341402 (N=99) | Non-switching: NovoLog (N=111)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Alcohol Abuse (Psychiatric disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switching: NovoLog/SAR341402 (N=99) | Non-switching: NovoLog (N=111)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT03874715/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT03874715/SAP_001.pdf